CLINICAL TRIAL: NCT00777114
Title: Phase 1 Study of Radiosensitization Using Bortezomib in Relapsed Non-Hodgkin's Lymphoma Patients Receiving Radioimmunotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0806009862; NCT00398762 (obsolete NCT alias)
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: relapsed non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bortezomib; tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental)
  Interventions: Drug: bortezomib, tositumomab

INTERVENTIONS:
Drug: bortezomib, tositumomab — 1. 0.30mg/m2 bortezomib and 50cGy 131I-tositumomab,
  2. 0.30 mg/m2 bortezomib and 75 cGy 131I-tositumomab,
  3. 0.60 mg/m2 bortezomib and 75 cGy 131I-tositumomab,
  4. 0.90 mg/m2 bortezomib and 75 cGy 131I-tositumomab, and
  5. 1.2 mg/m2 bortezomib and 75 cGy 131I-tositumomab.

SUMMARY:
This will be a multi-center, Phase I, dose-escalation study of bortezomib in combination with 131I-tositumomab in patients with relapsed non-Hodgkin's lymphoma. Bortezomib will be administered to patients twice weekly, with the first dose being given two days prior to the treatment dose of 131I-tositumomab, and the second dose two days after RIT for a total of 5 doses.

Patients will be enrolled and undergo standard staging studies, including history, physical examination, complete blood count, serum chemistries and LDH, TSH, HAMA, iliac crest bone marrow biopsy, and CT scans of the chest, abdomen and pelvis. All patients will provide written informed consent.

Bortezomib will be evaluated at 4 dose levels (0.30 mg/m2, 0.60 mg/m2, 0.90 mg/m2, and 1.2 mg/m2) and 131I-tositumomab at 2 dose levels (50 cGy and 75 cGy TBD). Bortezomib will be administrated the day prior to 131I-tositumomab and twice weekly thereafter for 4 doses in order to provide proteasome inhibition throughout the period of 131I-tositumomab activity. The intention is to use 131I-tositumomab at full dose if possible. Therefore, the 50cGy dose will be used only with the lowest dose of bortezomib in case of unexpected toxicities with the combination.

Dose levels will be as follow:

1. 0.30mg/m2 bortezomib and 50cGy 131I-tositumomab,
2. 0.30 mg/m2 bortezomib and 75 cGy 131I-tositumomab,
3. 0.60 mg/m2 bortezomib and 75 cGy 131I-tositumomab,
4. 0.90 mg/m2 bortezomib and 75 cGy 131I-tositumomab, and
5. 1.2 mg/m2 bortezomib and 75 cGy 131I-tositumomab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven relapsed or refractory MCL, DLBCL including subtypes mediastinal large B cell, centroblastic, immunoblastic, T cell rich B cell and anaplastic large B cell lymphoma, or low grade B cell NHL.
* Patients must have received prior systemic therapy for their lymphoma.
* Age >18 years.
* Life expectancy of greater than 12 weeks
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib or boron.
* Previous radiation therapy to the maximum tissue tolerance at any site.
* Previous autologous or allogeneic stem cell transplantation.
* Involvement of the bone marrow of >25% by lymphoma.
* Known involvement of the central nervous system by lymphoma. 17
* Significant organ dysfunction, including hematologic (absolute neutrophil count <1500, platelets <150,000).
* ECOG performance status >2.
* Uncontrolled illness including, but not limited to, ongoing or active infection,symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV infection.
* Patient has a calculated or measured creatinine clearance of <20 mL/minute within 14 days before enrollment.
* Patient has ≥Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 3 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2012-12-18 (Actual); Study Completion 2012-12-18 (Actual)

PRIMARY OUTCOMES:
The primary objectives of this study are to determine: a) The appropriate doses of bortezomib and 131I-tositumomab when used in combination. b) Toxicities of the combination treatment. | throughout dose escalation treatments

CONTACTS AND LOCATIONS:
Overall Officials: Jia Ruan, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medical College, New York, New York